CLINICAL TRIAL: NCT03684577
Title: Efficacy of Hypnotherapy Compared to a Wait-list Control Group in the Treatment of Agoraphobia
Brief Title: Efficacy of Hypnotherapy for Agoraphobia
Acronym: WIKI-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Anil Batra, Prof. Dr. Anil Batra, Pricinpal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WIKI-A
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Agoraphobia
Keywords: Hypnosis; Wait-list
MeSH Terms: conditions — Agoraphobia | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotherapy for Agoraphobia (Experimental): A total of 8-12 individual sessions of hypnotherapy over 12 weeks will be delivered. Hypnotherapy consists of hypnotic activation and reinforcement of the patient's own resources, the use of relevant positive and negative experiences from the biography, and the development of positive solution imagery. The central technique is the work with a symptom regression and the resolution of old and actual experiences. Furthermore, formal trance induction, utilisation techniques, indirect techniques such as the use of metaphors or the representative technique, or work with time progression will be used.
  Interventions: Behavioral: Hypnotherapy for Agoraphobia
- Wait-list control group (No Intervention): Patients in the wait-list control group will receive 8-12 sessions of individual hypnotherapy after a waiting period for 12 weeks.

INTERVENTIONS:
Behavioral: Hypnotherapy for Agoraphobia — see description of the experimental arm
  Arms: Hypnotherapy for Agoraphobia

SUMMARY:
The purpose of the study is to compare the efficacy of Hypnotherapy for the treatment of Agoraphobia compared to a wait-list control group.

DETAILED DESCRIPTION:
With the present study, the efficacy of 8-12 sessions of individual Hypnotherapy will be compared to a wait-list control groups. At study entry and at the end of treatment with Hypnotherapy, the Agoraphobia symptoms will be assessed via clinician-rating and self-report. It is expected that Hypnotherapy will be superior to a wait-list control regarding the percentage reduction of the anxiety symptoms after three months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patient fulfills DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria for agoraphobia
* 18 - 65 years of age
* Sufficient knowledge of the German language in order to participate in the study
* Sufficient availability to participate in weekly therapy sessions

Exclusion Criteria:

* Acute suicidality (intended action, concrete plans or intermittent pronounced suicidal ideation)
* Lifetime diagnosis of a bipolar disorder or psychotic disorder
* Alcohol or substance use disorder without abstinence in the last 12 months
* Severe cognitive impairments (in cases of suspicion evaluation via Mini Mental State Test (MMST) < 26, will be conducted)
* Other severe primary mental disorders to be treated: severe Major Depressive Disorder, severe personality disorder of borderline type with self-injury, severe combined personality disorder, actual posttraumatic stress disorder, anorexia nervosa, obsessive compulsive disorder
* Somatic disorder impeding participation in regular psychotherapy sessions
* Outpatient psychotherapy during the last twelve months.
* Medication with anxiolytics or anti-psychotics (antidepressant medication is permitted if stable since more than eight weeks and no planned changes during the duration of therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Panic and Agoraphobia Scale (PAS) | Between baseline (t1) and after 12 weeks (t2)
  The clinician-rating PAS will be used to measure the symptom severity (range 0-56 with higher values indicating more symptoms) for the primary outcome that is defined as the (mean) percentage change of the total symptom score between baseline (t1) and after 12 weeks (t2).

CONTACTS AND LOCATIONS:
Overall Officials: Anil Batra, Prof., Principal Investigator — University Hospital Tuebingen
Locations (1):
- Prof. Dr. A. Batra/ Dr. Kristina Fuhr, University Department for Psychiatry and Psychotherapie, Tübingen, Germany

REFERENCES:
- [Derived] Fuhr K, Bender A, Wiegand A, Janouch P, Drujan M, Cyrny B, Schweizer C, Kreifelts B, Nieratschker V, Batra A. Hypnotherapy for agoraphobia-Feasibility and efficacy investigated in a pilot study. Front Psychol. 2023 Aug 10;14:1213792. doi: 10.3389/fpsyg.2023.1213792. eCollection 2023. PMID 37637902